CLINICAL TRIAL: NCT04847375
Title: Evaluation of the Effect of Exogenous Surfactant Through Nebulizer Mask on Clinical Outcomes in Covid-19 Patients
Brief Title: Exogenous Surfactant Through Nebulizer Mask on Clinical Outcomes in Covid-19 Patients
Acronym: CovidSurf
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali Dabbagh, Clinical Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27348
Record Dates: First submitted 2021-04-10; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: COVID-19; Respiratory Distress Syndrome; Surface-Active Agents
Keywords: Covid-19; exogenous surfactant; Adult Respiratory Distress Syndrome; nebulizer
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor would be blind regarding the study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nebulized Surfactant (Experimental): The patients in this group will receive exogenous surfactant using nebulizer mask as soon as they are admitted in the hospital (ward or emergency department) with a diagnosis of COVID-19; in addition they will receive standard care based on the national guidelines
  Interventions: Drug: exogenous surfactant
- Standard Care (No Intervention): The patients in this group will receive standard care based on the national guidelines as soon as they are admitted in the hospital (ward or emergency department) with a diagnosis of COVID-19

INTERVENTIONS:
Drug: exogenous surfactant — Nebulized Surfactant would be administered by face mask which has a nebulizer
  Arms: Nebulized Surfactant

SUMMARY:
Covid-19 disease is one of the most important health system challenges which is the result of the recent SARS CoV-2 virus outbreak. So far, despite the use of different types of pharmaceuticals, none has been served as a curative treatment and research is continued to find one or more effective drugs; either palliative or curative ones.

One of the most important clinical problems in Covid-19 patients is lung involvement, which may causes significant sequels; leading to a main part of morbidity and/or mortality.

Surfactant is one of the drugs that can have valuable effects on the lungs, both by reducing the alveolar surface tension and by exerting immunomodulatory effects.

In a previous study by the same team, favorable effects were seen in intubated patients; however, the aim of this study was to evaluate the effect of exogenous nebulized surfactant in the pre-intubation stages of the disease.

DETAILED DESCRIPTION:
Exogenous surfactant in neonates with clinical pulmonary distress syndrome has demonstrated pulmonary improvement; the latter being one of the most important applications of exogenous surfactant. In adults with underlying lung disease, especially Adult Respiratory Distress Syndrome (ARDS), there are controversial findings regarding the efficacy of surfactant.

However, in a previous study, it was shown that surfactant in COVID-19 patients with pulmonary intubation improved pulmonary function and gas exchange and also, reduced patient mortality.

However, none of the other repurposed drugs in COVID-19 have yet been able to prove significant effects in the treatment of patients; based on a recent study on more than 11000 COVID-19 patients (i.e. the SOLIDARITY study).

Due to the significant worldwide challnege with COVID-19, many efforts have been made in this regard, but the definitive cure has not yet been obtained, and therefore, efforts are being made to find an effective method to treat the disease and improve patients' symptoms; parallel to the efforts to increase the vaccination coverage.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* definitive proof of COVID-19 infection by polymerase chain reaction (PCR) within 48 hours of hospital admission
* COVID-19 related Moderate ARDS following Berlin criteria definition with PaO2/FiO2 < 200 requiring what condition?
* Signed and dated informed consent form (ICF) by the subject or caregivers

Exclusion Criteria:

* known or high suspicion of pre-existing heart failure, unstable angina
* presence of severe shock with hemodynamic instability despite escalating vasopressors
* Severe, underlying pulmonary infection or severe pulmonary disease except for COVID-19 (COPD, pulmonary fibrosis, lung cancer, bacterial pneumonia, etc.)
* Diagnosis of pulmonary hemorrhage
* Pregnancy or lactation
* Other significant cause than ARDS to the respiratory failure
* Age less than 18
* Age more than 80
* Need for ECMO (extracorporeal membrane oxygenation) during the study
* Anticipated transfer to another hospital within 72 hours
* Known hypersensitivity to exogenous surfactant
* Current participation or participation in another study within the last month that in the opinion of the investigator would prevent enrollment for safety purposes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-20 (Estimated); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
rate of tracheal intubation | through study completion, an average of 1 year
  the frequency of patients who will be intubated due to deteriorated pulmonary function
rate of ICU admission | through study completion, an average of 1 year
  the frequency of patients who will be admitted to intensive care unit due to deteriorated pulmonary function
lowest oxygen saturation | through study completion, an average of 1 year
  lowest number reading in the pulse oxymetry in one of the fingers or toes

SECONDARY OUTCOMES:
30 days mortality | the first 30 days after hospital admission
  the mortality rate during the first 30 days after the first day of hospital admission
90 days mortality | the first 90 days after hospital admission
  the mortality rate during the first 90 days after the first day of hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Zarghi, PhD, Study Chair — Deputy of Research and Technology, Shahid Beheshti University of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided
to be determined

REFERENCES:
- [Background] Ghahremani M, Fathi M, Massoudi N, Tavana S, Fani K, Nooraee N, Malekpour Alamdari N, Besharat S, Naja Abrandabadi A, Pirsalehi A, Khabiri Khatiri MA, Amini Pouya M, Rajaei S, Dabbagh A. Exogenous Surfactant Versus Placebo in the Treatment of Moderate and Severe ARDS in COVID19: The Pilot Study of a Clinical Trial. DOI: https://doi.org/10.21203/rs.3.rs-136365/v1. Preprint.
- [Result] Takian A, Raoofi A, Kazempour-Ardebili S. COVID-19 battle during the toughest sanctions against Iran. Lancet. 2020 Mar 28;395(10229):1035-1036. doi: 10.1016/S0140-6736(20)30668-1. Epub 2020 Mar 18. No abstract available. PMID 32199073
- [Result] Zhang Y, Xu J, Li H, Cao B. A Novel Coronavirus (COVID-19) Outbreak: A Call for Action. Chest. 2020 Apr;157(4):e99-e101. doi: 10.1016/j.chest.2020.02.014. Epub 2020 Feb 19. No abstract available. PMID 32087216
- [Result] Yue H, Bai X, Wang J, Yu Q, Liu W, Pu J, Wang X, Hu J, Xu D, Li X, Kang N, Li L, Lu W, Feng T, Ding L, Li X, Qi X; Gansu Provincial Medical Treatment Expert Group of COVID-19. Clinical characteristics of coronavirus disease 2019 in Gansu province, China. Ann Palliat Med. 2020 Jul;9(4):1404-1412. doi: 10.21037/apm-20-887. Epub 2020 Jul 13. PMID 32692208
- [Result] INSPIRATION Investigators; Sadeghipour P, Talasaz AH, Rashidi F, Sharif-Kashani B, Beigmohammadi MT, Farrokhpour M, Sezavar SH, Payandemehr P, Dabbagh A, Moghadam KG, Jamalkhani S, Khalili H, Yadollahzadeh M, Riahi T, Rezaeifar P, Tahamtan O, Matin S, Abedini A, Lookzadeh S, Rahmani H, Zoghi E, Mohammadi K, Sadeghipour P, Abri H, Tabrizi S, Mousavian SM, Shahmirzaei S, Bakhshandeh H, Amin A, Rafiee F, Baghizadeh E, Mohebbi B, Parhizgar SE, Aliannejad R, Eslami V, Kashefizadeh A, Kakavand H, Hosseini SH, Shafaghi S, Ghazi SF, Najafi A, Jimenez D, Gupta A, Madhavan MV, Sethi SS, Parikh SA, Monreal M, Hadavand N, Hajighasemi A, Maleki M, Sadeghian S, Piazza G, Kirtane AJ, Van Tassell BW, Dobesh PP, Stone GW, Lip GYH, Krumholz HM, Goldhaber SZ, Bikdeli B. Effect of Intermediate-Dose vs Standard-Dose Prophylactic Anticoagulation on Thrombotic Events, Extracorporeal Membrane Oxygenation Treatment, or Mortality Among Patients With COVID-19 Admitted to the Intensive Care Unit: The INSPIRATION Randomized Clinical Trial. JAMA. 2021 Apr 27;325(16):1620-1630. doi: 10.1001/jama.2021.4152. PMID 33734299
- [Result] Dabbagh A, Rajaei S, Ghahremani M, Fathi M, Massoudi N, Tavana S, Fani K, Nooraee N, Malekpour Alamdari N, Besharat S, Najafi Abrandabadi A, Pirsalehi A, Khabiri Khatiri MA. The effect of surfactant on clinical outcome of patients with COVID-19 under mechanical ventilation: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Nov 11;21(1):919. doi: 10.1186/s13063-020-04815-z. PMID 33176850
- [Result] Alamdari NM, Afaghi S, Rahimi FS, Tarki FE, Tavana S, Zali A, Fathi M, Besharat S, Bagheri L, Pourmotahari F, Irvani SSN, Dabbagh A, Mousavi SA. Mortality Risk Factors among Hospitalized COVID-19 Patients in a Major Referral Center in Iran. Tohoku J Exp Med. 2020 Sep;252(1):73-84. doi: 10.1620/tjem.252.73. PMID 32908083
- [Result] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846